CLINICAL TRIAL: NCT05644678
Title: Comparison of Posttreatment Periodontal Status of Palatally Impacted Canines Aligned by Conventional Versus Accelerated Minimally-invasive Corticotomy-assisted Orthodontic Traction Treatment: A Randomized Controlled Trial
Brief Title: Evaluation of the Periodontal Status After the Treatment of Palatally Impacted Canines Using Acceleration Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-15-2022
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Impacted Canine
Keywords: Impacted canine; accelerate canine traction; periodontal index; periodontal status
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Patients will be treated using the fixed appliances to track the impacted canines after opening the appropriate distance
  Interventions: Device: Fixed appliances
- Surgically-assisted treatment (Experimental): Patients will be treated using fixed appliances assisted by minimally-invasive corticotomy (alveolar perforations and piezocision) to accelerate impacted canines' traction after opening the appropriate distance.
  Interventions: Procedure: Corticotomy

INTERVENTIONS:
Device: Fixed appliances — Metal brackets with a straight-wire prescription will be used. Patients will be treated conventionally.
  Arms: Conventional treatment
Procedure: Corticotomy — Patients will be treated in conjunction with a surgical intervention using metal brackets with a straight-wire prescription. Corticotomy (alveolar perforation and piezocision) will induce acceleration in canine traction movement during the orthodontic treatment in only one group.
  Arms: Surgically-assisted treatment

SUMMARY:
Impacted canine causes many problems for patients, such as damage to the adjacent teeth roots, effects on gingival tissues, aesthetic problems, difficulty, and prolonged orthodontic treatment duration. Therefore, solutions to accelerate the movement of impacted canines with the help of surgical procedures to reduce treatment time will be investigated, such as intra-operative alveolar perforations and piezocision. We also aimed to evaluate periodontal changes associated with such accelerating procedures compared with the conventional traction method.

DETAILED DESCRIPTION:
Patients with palatally impacted maxillary canines will be treated using fixed appliances assisted by some surgical procedures. The effects of this treatment approach on the periodontal status will be assessed using periodontal measurements.

There are two groups :

1. conventional treatment group
2. minimally-invasive corticotomy-assisted treatment group Patients will be allocated to the two groups randomly. Data will be collected using periodontal variables.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients: 18-28 years.
2. Palatal or Mid-alveolar impacted canine.
3. There is no previous orthodontic treatment.
4. Healthy periodontal tissues and good oral health (i.e., the Plaque Index is less or equal to 1 according to Loe and Silness(1963).
5. The patient does not take any drug that may interfere with the tooth movement (Cortisone, NSAIDs …).
6. Mild or no crowding on the upper jaw.
7. No history of previous trauma to the maxillofacial region or surgical interventions.

Exclusion Criteria:

1. Any systemic diseases that would affect tooth movement
2. Antidepressant prevents oral surgery
3. Any congenital syndromes or cleft lip and palate cases
4. Bad oral health
5. Previous orthodontic treatment

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in the periodontal pocket depth (PPD) | Time 1: immediately before the surgical exposure; Time 2: immediately at the end of the active treatment
  The distance from the gingival margin to the base of the pocket of the first premolar, canine, and lateral incisor.
Changes in the gingival margin (GM) | Time 1: immediately before the surgical exposure; Time 2: immediately at the end of the active treatment
  The distance from the cementoenamel junction (CEJ) to the gingival margin of the first premolar, canine, and lateral incisor.
Changes in the width of the keratinized tissue (KT) | Time 1: immediately before the surgical exposure; Time 2: immediately at the end of the active treatment
  The distance from the gingival margin to the mucogingival junction of the first premolar, canine, and lateral incisor

SECONDARY OUTCOMES:
Changes in the Gingival Index (GI) | Time 1: immediately before the surgical exposure; Time 2: immediately at the end of the active treatment
  The gingival status will be assessed using the following classification 0= Normal gingiva.
  1. Mild inflammation: slight color change, slight edema, No bleeding on probing.
  2. Moderate inflammation: redness, edema and glazing. Bleeding on probing.
  3. Severe inflammation: marked redness and edema. Tendency to spontaneous bleeding. Ulceration.
Changes in the Bleeding Index (BI) | Time 1: immediately before the surgical exposure; Time 2: immediately at the end of the active treatment
  The healthiness of the gingival margin and the attached gingivae will be assessed depending on the status of gingival inflammation.
  0= No bleeding.
  1. Bleeding some seconds after probing.
  2. Bleeding immediately after probing.
  3. Bleeding on probing spreading towards the marginal gingiva.

CONTACTS AND LOCATIONS:
Overall Officials: Mahran R Mousa, DDS,MSc, Study Chair — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria; Omar Heshmeh, DDS,MSc,PhD, Study Director — Department of oral and maxillofacial surgery, Damascus University, Syriam
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smailiene D, Kavaliauskiene A, Pacauskiene I, Zasciurinskiene E, Bjerklin K. Palatally impacted maxillary canines: choice of surgical-orthodontic treatment method does not influence post-treatment periodontal status. A controlled prospective study. Eur J Orthod. 2013 Dec;35(6):803-10. doi: 10.1093/ejo/cjs102. Epub 2013 Jan 24. PMID 23349422
- [Background] Parkin NA, Milner RS, Deery C, Tinsley D, Smith AM, Germain P, Freeman JV, Bell SJ, Benson PE. Periodontal health of palatally displaced canines treated with open or closed surgical technique: a multicenter, randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):176-84. doi: 10.1016/j.ajodo.2013.03.016. PMID 23910198
- [Background] Crescini A, Nieri M, Buti J, Baccetti T, Mauro S, Prato GP. Short- and long-term periodontal evaluation of impacted canines treated with a closed surgical-orthodontic approach. J Clin Periodontol. 2007 Mar;34(3):232-42. doi: 10.1111/j.1600-051X.2006.01042.x. Epub 2007 Jan 25. PMID 17257160
- [Background] Pini Prato G, Baccetti T, Magnani C, Agudio G, Cortellini P. Mucogingival interceptive surgery of buccally-erupted premolars in patients scheduled for orthodontic treatment. I. A 7-year longitudinal study. J Periodontol. 2000 Feb;71(2):172-81. doi: 10.1902/jop.2000.71.2.172. PMID 10711607
- [Background] Crescini A, Clauser C, Giorgetti R, Cortellini P, Pini Prato GP. Tunnel traction of infraosseous impacted maxillary canines. A three-year periodontal follow-up. Am J Orthod Dentofacial Orthop. 1994 Jan;105(1):61-72. doi: 10.1016/S0889-5406(94)70100-8. PMID 8291494
- [Background] Zasciurinskiene E, Bjerklin K, Smailiene D, Sidlauskas A, Puisys A. Initial vertical and horizontal position of palatally impacted maxillary canine and effect on periodontal status following surgical-orthodontic treatment. Angle Orthod. 2008 Mar;78(2):275-80. doi: 10.2319/010907-8.1. PMID 18251594